CLINICAL TRIAL: NCT00581893
Title: Phenytoin and Driving Safety: A Randomized, Controlled Cross-Over Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Erik St. Louis, Assistant Professor (Clinical), University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 200512712; 5R49CE721682-05 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cognitive Measures; Driving Simulator Performance
Keywords: epilepsy; cognitive impairment; driving simulation; cross-over study
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction | interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Phenytoin administration
  Interventions: Drug: Phenytoin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Phenytoin — Phenytoin will be dosed to a target dose of 5 mg/kg qhs for one month
  Other Names: Dilantin
  Arms: 1
Drug: Placebo oral capsule — Placebo
  Arms: 2

SUMMARY:
Automobile driving is a crucial aspect of everyday life, yet vehicular crashes represent a serious public health problem. Patients with epilepsy are at elevated risk for automobile crashes, causing great personal suffering and financial costs to society. Most collisions involving epileptic drivers are not seizure related but may instead result from cognitive effects upon driving performance of epilepsy and antiepileptic drugs (AEDs). Several million American drivers take AEDs for treatment of medical conditions besides epilepsy and may also be at risk for cognitive impairments that can reduce driving performance. Empirical evidence of the effects of AEDs on driving performance would enable development of driving guidelines that could lower the risk of injurious motor vehicle collisions; however, this evidence is currently lacking. The broad goal of our project is to determine the specific effects of the most commonly utilized AED, phenytoin, by assessing driving performance and cognitive abilities in neurologically normal volunteers taking phenytoin in a randomized, double-blind, placebo-controlled, crossover study. Our proposed experiments will assess: (1) cognitive functions using standardized neuropsychological tests (of attention, perception, memory, and executive functions), (2) driving performance during phenytoin and placebo administration, and (3) the effects of phenytoin-related cognitive performance upon driving performance. To measure driving performance, we will use a state-of-the-art fixed-base interactive driving simulator that allows us to observe driver errors in an environment that is challenging yet safe for the driver and tester, under conditions of optimal stimulus and response control. The results of this study of 30 drivers treated with phenytoin and placebo will increase the understanding of the role of AED-related cognitive impairment on driving safety errors. A better understanding of the impact of AEDs upon driving performance is necessary to rationally develop interventions that could help prevent crashes by drivers treated with AEDs.

DETAILED DESCRIPTION:
Patients with epilepsy are at elevated risk for automobile crashes, causing great personal suffering and financial costs to society. Most collisions involving epileptic drivers are not seizure related but may instead result from cognitive effects upon driving performance of epilepsy and antiepileptic drugs (AEDs). Several million American drivers take AEDs for treatment of medical conditions besides epilepsy and may also be at risk for cognitive impairments that can reduce driving performance. Empirical evidence of the effects of AEDs on driving performance would enable development of driving guidelines that could lower the risk of injurious motor vehicle collisions; however, this evidence is currently lacking.

The broad goal of the current project is to determine the specific effects of AEDs on cognitive function and driving performance. To address this goal we will assess driving performance and cognitive abilities in neurologically normal volunteers taking phenytoin (Dilantin), the most commonly prescribed AED. Effects of phenytoin on driving performance and cognition will be addressed in a randomized, double-blind, placebo-controlled, crossover study. Driver cognition will be assessed using a battery of neuropsychological tests. Driving performance will be objectively assessed in all participants on standardized tasks enacted in a state-of-the-art driving simulator. Our 3 Specific Aims are:

Aim 1: To assess the effects of phenytoin on cognitive abilities that are crucial to the driving task, including perception, attention, memory, and executive function.

Hypothesis 1: A driver's cognitive abilities will decline during steady-state phenytoin administration compared to placebo. Drivers with higher blood levels of phenytoin will show greater decline.

Aim 2: To assess effects of phenytoin on driving performance and safety errors in a state-of-the-art driving simulator.

Hypothesis 2: Driving performance will decline and driver safety errors will increase during phenytoin administration compared to placebo. Drivers with higher blood levels of phenytoin will show greater impairments of driving.

Aim 3: To assess the effects of phenytoin-related cognitive impairments upon driving performance in a state-of-the-art driving simulator.

Hypothesis 3. Impairments of cognitive function affecting perception, attention, memory, executive function, and arousal will increase the likelihood of driver errors that may lead to a crash.

Our hypotheses would be supported if the drivers taking phenytoin, as opposed to placebo, demonstrate worse cognitive performance on neuropsychological tests, and more safety errors and crashes in the simulator. The hypotheses would also be supported if drivers with higher phenytoin levels show greater impairments of cognition and driving. Once the effects of phenytoin on driving performance are demonstrated in this project, we will have evidence to support more comprehensive research addressing specific dosing and serum levels and acute versus chronic administration.

There is currently no evidence concerning the effects of phenytoin on driving performance. Accurate driving performance data on patients receiving phenytoin would allow determination of fair and accurate criteria for making recommendations to drive or not to drive affecting millions of patients taking AEDS for epilepsy and other conditions. These data could also help reduce the risk of car crashes due to medication side effects.

ELIGIBILITY:
Inclusion Criteria:

* Anticipating a 10-15% drop-out rate, we will induct 30 neurologically normal subjects (age 18 (21) -60) to obtain 25 evaluable subjects who are legally licensed to drive in their state of residence and have been actively driving under appropriate legal guidelines for at least 5 years (to minimize performance variations of novice drivers).
* Because this study is intended to determine the potential effects of phenytoin on driving performance, a relatively healthy cohort of patients must be chosen. Chronic medical or psychiatric conditions could cause significant alterations in driving performance independent of those caused by phenytoin, which would complicate interpretation of performance impairments.

Exclusion Criteria:

* Subjects who are younger than 18 or older than 60
* Have history of prior seizures, family history of epilepsy, or prior history of head injury
* Have a known history of prior drug or alcohol abuse or unwillingness to abstain from drug or alcohol use during the study period
* Have a past or current active neurological or psychiatric disorder that could impair cognitive or driving performance (i.e. baseline IQ < 90, dementia, mental retardation, stroke, severe head injury, schizophrenia, active clinical depression, progressive brain tumor).
* Subjects who have a chronic medical condition (i.e. diabetes mellitus, renal insufficiency, congestive heart failure, hepatic dysfunction, hematologic condition, HIV)
* Taking medications known to affect the central nervous system (i.e. baseline pre-study treatment with antiepileptic drug, anxiolytics, sedatives, hypnotics, antidepressants, antipsychotics, narcotics and tranquilizers)
* Regularly use over-the-counter cough suppressants, antihistamines, or sleep aids; or who ingest over 7 cups of daily coffee or currently smoke cigarettes.
* Subjects will be excluded if they cannot complete SIREN testing or neuropsychological instruments because of visual or hearing impairment (history or screening discovery of corrected visual acuity of less than 20/50) or other physical disability, or if they have a history of severe motion sickness as an adult-a marker for patients who develop simulator sickness and therefore cannot participate in SIREN testing.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik K St. Louis, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] St. Louis EK, McEvoy S, Shi QC, Rizzo M. Useful Field of View impairment in partial epilepsy. Unpublished observations and submitted abstract to 3rd International Driving Symposium on Human Factors in Driving Asssessment, Training, and Vehicle Design, Rockport, Maine, June, 2005.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phenytoin First, Then Placebo: Subjects first received Phenytoin target dose of 5 mg/kg qhs for one month. After a 14 day washout period, they received the placebo treatment for one month.
- Placebo First, Then Phentoin: Subjects first received Placebo for one month. After a 14 day washout period, they received Phenytoin target dose of 5 mg/kg qhs for one month.
Period: First Intervention (1 Month)
Arm/Group | Phenytoin First, Then Placebo | Placebo First, Then Phentoin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Phenytoin First, Then Placebo | Placebo First, Then Phentoin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Second Intervention (1 Month)
Arm/Group | Phenytoin First, Then Placebo | Placebo First, Then Phentoin
Started | 10 | 10
Completed | 7 | 8
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cross-over Design: Subjects will be studied on two occasions, in random order. They will randomly be assigned to received either Phenytoin target dose of 5 mg/kg qhs for one month or placebo treatment for one month. After a 14 day washout period, they will receive the opposite treatment from the original.
Arm/Group | Cross-over Design
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had a Driving Simulator Crash Event
Description: Number of subjects who had a crash event during the driving simulator test.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Groups:
- Phenytoin: Phenytoin target dose of 5 mg/kg
- Placebo: Placebo oral capsule
Arm/Group | Phenytoin | Placebo
Number analyzed (Participants) | 20 | 20
Participants | 2 | 0
Statistical Analysis 1: Comparison: Phenytoin vs Placebo; Test type: Superiority; p = 0.50, McNemar

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study, approximately 2.5 months, for an overall duration of approximately three years.
Groups:
- Phenytoin: Phenytoin target dose of 5 mg/kg qhs
Arm/Group | Phenytoin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
The very small sample size of evaluable subjects prevents definitive conclusions on the safety hazards of phenytoin for driving performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes